CLINICAL TRIAL: NCT04730739
Title: FastFrame™ External Fixation System Post-Market Clinical Follow-Up Study: Knee Spanning Kit and Damage Control Kit
Brief Title: FastFrame Knee Spanning and Damage Control Kit PMCF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product will not be taken to EU, thus no PMCF requirements.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMU2017-95T
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Fracture; Fractures, Bone; Fractures, Closed; Fractures, Open
Keywords: External fixator, temporary stabilization
MeSH Terms: conditions — Fractures, Bone; Fractures, Closed; Fractures, Open

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FastFrame External Fixation System - Knee Spanning or Damage Control Kit (Experimental): The patient must have been treated with either Knee Spanning or Damage Control FastFrame External Fixation System.
  Interventions: Device: FastFrame External Fixation System - Knee Spanning or Damage Control Kit

INTERVENTIONS:
Device: FastFrame External Fixation System - Knee Spanning or Damage Control Kit — The FastFrame External Fixation Systems - Knee Spanning Kit and Damage Control Kit are single-use external fixators that are sterile packed with all required components for convenience of the end user.

SUMMARY:
The purpose of this prospective study is to confirm safety and performance of the FastFrame External Fixation System and corresponding instrumentation.

DETAILED DESCRIPTION:
Study Title: FastFrame™ External Fixation System Post-Market Clinical Follow-Up Study (Knee Spanning Kit and Damage Control Kit)

Sponsor: Zimmer Biomet

Study Design: Prospective enrollment, prospective follow-up, single cohort study

Clinical Phase: Postmarket

Number of Sites: Up to three sites

Study Duration per Subject: Subjects will be enrolled in the study until the time of exchange of their FastFrame Kit to another device. Typically, this exchange occurs 2-4 weeks after injury.

Primary Objective: The objective of this observational, prospective study is to confirm safety and performance of the FastFrame External Fixation System and corresponding instrumentation.

Primary Endpoint: Frequency and incidence of device-related adverse events and device deficiencies before the FastFrame External Fixation System is exchanged by another device (i.e. plates, screws, etc.).

Secondary Endpoint: Adverse events that occur between application of the FastFrame External Fixation System and exchange with another device that do not fall within the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older
* Patient must be treated with either the Knee Spanning or Damage Control FastFrame External Fixation System according to the European Economic Area (EEA) indications*

EEA Indications (a subset of the cleared US indications):

The FastFrame External Fixation System - Knee Spanning Kit is indicated for use in treatment of long bone (distal femur, proximal tibia) fractures. Specifically, the system is intended for temporary stabilization of open or closed fractures about the knee, typically in the context of polytrauma or where open or alternative closed treatment is undesirable or otherwise contraindicated.

The FastFrame External Fixation System - Damage Control Kit is indicated for use in treatment of mid-shaft long bone (femur, tibia) fractures. Specifically, the system is intended for temporary stabilization of open or closed fractures of the femur and tibia, typically in the context of polytrauma or where open or alternative closed treatment is undesirable or otherwise contraindicated.

Exclusion Criteria:

* Patient has an active or suspected infection
* Patient has conditions that limit their ability and/or willingness to follow instructions during the healing process
* Patient has inadequate skin, bone, or neurovascular status
* Patient is a prisoner
* Patient is pregnant and/or breastfeeding
* Patient is a known current alcohol and/or drug abuser in the opinion of the Investigator
* Patient has a mental or neurologic condition that will not allow for proper Informed Consent and/or participation in follow-up program in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FastFrame External Fixation System - Knee Spanning or Damage Control Kit
Started | 33
Completed | 32
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | FastFrame External Fixation System - Knee Spanning or Damage Control Kit
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 49.28 [20 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device-related Adverse Events and Device Deficiencies
Description: Frequency and incidence of device-related adverse events and device deficiencies before the FastFrame External Fixation System is exchanged by another device (i.e. plates, screws, etc.).
Time Frame: 2-4 weeks postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | FastFrame External Fixation System - Knee Spanning or Damage Control Kit
Number analyzed (Participants) | 33
Participants | 0

2. Secondary Outcome: Number of Participants With Another Device-related Adverse Events
Description: Adverse events that occur between application of the FastFrame External Fixation System and exchange with another device that do not fall within the primary endpoint.
Time Frame: 2-4 weeks postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | FastFrame External Fixation System - Knee Spanning or Damage Control Kit
Number analyzed (Participants) | 33
Participants | 2

ADVERSE EVENTS:
Time Frame: Per the protocol, International Organization for Standardization (ISO) definitions were followed for adverse event data collection. All adverse events were captured for subjects enrolled through 2 - 4 weeks follow-up or study completion (including lost to follow-up), whichever came first.
Description: ISO definition is not materially different from clinicaltrials.gov definitions.
Arm/Group | FastFrame External Fixation System - Knee Spanning or Damage Control Kit
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FastFrame External Fixation System - Knee Spanning or Damage Control Kit (N=33)
Not Related (Musculoskeletal and connective tissue disorders) | 1 — BELOW KNEE AMPUTATION FOR DEVITALIZED TISSUES AND EXTENSIVE INJURY TO LEFT KNEE.
Not Related (Infections and infestations) | 1 — MAJOR COMPLICATIONS OR COMORBIDITIES COMPLICATED BY INVASIVE FUNGAL INFECTION IN ABDOMEN WITH SUBSEQUENT ISCHEMIC BOWEL, SEPSIS, AND DEATH. NO INFECTION PRESENT AT FRACTURE SITE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT04730739/Prot_SAP_000.pdf